CLINICAL TRIAL: NCT00136760
Title: Incentives Plus Bupropion for Smoking in Schizophrenics
Brief Title: Contingent Incentives Plus Bupropion for Smoking in People With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Tidey, Associate Professor (Research), Dept Psychiatry and Human Behavior, Brown University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-17566-1; R01DA017566 (NIH); R01-17566-1
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Tobacco Use Disorder
Keywords: tobacco
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Contingent reinforcement plus bupropion
  Interventions: Drug: Bupropion
- 2 (Experimental): Contingent reinforcement plus placebo
  Interventions: Drug: Contingent reinforcement plus placebo
- 3 (Experimental): Non-contingent reinforcement plus bupropion
  Interventions: Drug: non-contingent reinforcement plus bupropion
- 4 (Placebo Comparator): Non-contingent reinforcement plus placebo
  Interventions: Drug: Non-contingent reinforcement plus placebo

INTERVENTIONS:
Drug: Bupropion — Contingent reinforcement plus bupropion (300 mg/day for 3 weeks)
  Other Names: zyban, wellbutrin
  Arms: 1
Drug: Contingent reinforcement plus placebo — contingent reinforcement plus placebo (3 weeks)
  Arms: 2
Drug: non-contingent reinforcement plus bupropion — non-contingent reinforcement plus bupropion (300 mg/day for 3 weeks)
  Other Names: zyban, wellbutrin
  Arms: 3
Drug: Non-contingent reinforcement plus placebo — Non-contingent reinforcement plus placebo
  Arms: 4

SUMMARY:
There is a high prevalence of smoking among people with schizophrenia, and there are few smoking treatment programs for these smokers. The aims of this study are to investigate the separate and combined effects of bupropion and a voucher incentive program on smoking in people with schizophrenia.

DETAILED DESCRIPTION:
There is a high prevalence of smoking among people with schizophrenia, and there are few smoking treatment programs for these smokers. In this study, we are investigating whether the combination of bupropion (also called Zyban and Wellbutrin) and a behavioral treatment program (contingent vouchers) can reduce smoking in people with schizophrenia. This is a 3-week study aimed to investigate the feasibility of this treatment approach. Participants are randomly assigned to bupropion (300 mg/day, in 2 divided doses) or placebo. After one week on medication, participants are randomly assigned to the active behavioral treatment (contingent vouchers) or the control treatment (non-contingent vouchers). Over a 3-week period, participants come to the study site about 2-3 times per week, and provide information about their recent smoking and nicotine withdrawal symptoms. They also give saliva and urine samples that are analyzed for levels of cotinine, a nicotine metabolite. Participants in the active behavioral treatment group receive gift cards to local grocery stores when their cotinine levels indicate that they have reduced their smoking. Participants in the control behavioral treatment group receive gift cards regardless of cotinine level. Any participant who significantly reduces their smoking at the end of the trial is followed up 2 and 4 weeks after the end of the trial too see if they have sustained these smoking reductions. If we have favorable results from this trial, we will expand it into a smoking treatment program.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of schizophrenia or schizoaffective disorder, smoke 20-50 cpd, clinically stable on antipsychotic and antidepressant medications

Exclusion Criteria:

Pregnant/nursing women, seizure disorder, lowered seizure threshold due to other medical conditions, positive urine drug screen positive breath alcohol test, past 2 weeks use of MAO inhibitors, any form of bupropion, cimetidine, phenobarbital, phenytoin, DA agonists, anorectics, stimulants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W. Tidey, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Result] Tidey JW, Rohsenow DJ, Kaplan GB, Swift RM, Reid N. Effects of contingency management and bupropion on cigarette smoking in smokers with schizophrenia. Psychopharmacology (Berl). 2011 Sep;217(2):279-87. doi: 10.1007/s00213-011-2282-8. Epub 2011 Apr 8. PMID 21475970
- [Result] Tidey JW. Using incentives to reduce substance use and other health risk behaviors among people with serious mental illness. Prev Med. 2012 Nov;55 Suppl(Suppl):S54-60. doi: 10.1016/j.ypmed.2011.11.010. Epub 2011 Dec 9. PMID 22197799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community, using advertisements, and were recruited from an outpatient clinic at a local VA medical Center.
Pre-assignment Details: Participants underwent telephone and in-person screening for eligibility criteria.
Groups:
- CM + BUP: Contingent reinforcement plus bupropion
- CM + PLA: Contingent reinforcement plus placebo
- NR + BUP: Non-contingent reinforcement plus bupropion
- NR + PLA: Non-contingent reinforcement plus placebo
Period: Overall Study
Arm/Group | CM + BUP | CM + PLA | NR + BUP | NR + PLA
Started | 12 | 16 | 11 | 13
Completed | 12 | 16 | 11 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CM + BUP | CM + PLA | NR + BUP | NR + PLA | Total
Number analyzed (Participants) | 12 | 16 | 11 | 13 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 10 | 13 | 47
  >=65 years | 0 | 4 | 1 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.9) | 46.3 (6.7) | 43.7 (7.3) | 46.9 (6.8) | 45.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 2 | 15
  Male | 8 | 10 | 8 | 11 | 37
Region of Enrollment [Number; unit: participants]
  United States | 12 | 16 | 11 | 13 | 52

OUTCOME MEASURES:

1. Primary Outcome: Urinary Cotinine
Description: Urinary Cotinine levels at Week 4 (average of last 3 study visits)
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CM + BUP | CM + PLA | NR + BUP | NR + PLA
Number analyzed (Participants) | 12 | 16 | 11 | 13
ng/ml | 755 (533) | 1102 (639) | 1534 (489) | 1408 (490)

2. Secondary Outcome: Cigarettes Smoked Per Day
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | CM + BUP | CM + PLA | NR + BUP | NR + PLA
Number analyzed (Participants) | 12 | 16 | 11 | 13
cigarettes per day | 12.7 (7.4) | 13.9 (9.5) | 18.8 (12.9) | 21.0 (9.3)

ADVERSE EVENTS:
Arm/Group | CM + BUP | CM + PLA | NR + BUP | NR + PLA
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 4/12 | 0/16 | 3/11 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CM + BUP (N=12) | CM + PLA (N=16) | NR + BUP (N=11) | NR + PLA (N=13)
opiate detoxification (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — self-report
diarrhea, vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — self-report
fall (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blackout (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — self-report, not related
anxiety, restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — self-report, not related
bleeding ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — self-report, not related
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — self-report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes